CLINICAL TRIAL: NCT02855515
Title: The Role of Drug-Induced Sleep Endoscopy for the Optimisation of Treatment of Patients With Obstruction Sleep Apnoea
Brief Title: Drug-Induced Sleep Endoscopy for the Optimisation of Treatment of Patients With Obstruction Sleep Apnoea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FNO-ENT-DISE
Record Dates: First submitted 2016-07-26; First posted 2016-08-04 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Obstructive Sleep Apnoea; Sleep-Disordered Breathing
Keywords: drug-induced sleep endoscopy; obstructive sleep apnoea; VOTE classification; AHI; BMI
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Short-time diagnostic anaesthesia (Experimental): The study population will consist of patients with obstructive sleep apnoea, which will be classified as mild, moderate, severe (patients who failed or refused primary CPAP treatment). The patients will undergo a short-time general anaesthesia in order to diagnose OSA when relaxed.
  Interventions: Procedure: Short-time diagnostic anaesthesia

INTERVENTIONS:
Procedure: Short-time diagnostic anaesthesia — Patients will undergo a short-time general anaesthesia in order to diagnose Obstructive Sleep Apnoea when relaxed.

SUMMARY:
The main diagnostic challenge in patients with OSA (obstructive sleep apnea) is to determine the location of obstruction of the upper airway during sleep. This is so, because the otorhinolaryngology examination, which states probable site of obstruction of upper airways, is performed in the awake status. Therefore, drug-induced sleep endoscopy (DISE) has been introduced in the diagnostic algorithm of OSA patients during the last decade. The advantage of DISE is, that the collapse of upper airways, which is not visible during the awake status can be observed and targeted therapy according to the location and degree of obstruction of the upper airway can be applied. As a result, higher treatment success in patients with OSA can be reached.

DETAILED DESCRIPTION:
Materials and Methods The study was approved by the Institutional Ethics Committee and performed in accordance with the Declaration of Helsinki, good clinical practice, and applicable regulatory requirements. Informed written consent was obtained from all participants before initiation of any procedure.

• History, otorhinolaryngology examination, polysomnography Patient history will be taken with emphasis on snoring and OSA symptoms. Daytime sleepiness will be assessed using the Epworth Sleepiness Scale. Moreover, patients will be asked to grade the severity of snoring on a 10-point Visual Analogue Scale (0 = no snoring, 10 = extreme snoring). The body mass index (BMI) will be calculated.

Otorhinolaryngology examination, focusing on nasal, pharyngeal and laryngeal pathologies (enlargement of uvula, soft palate webbing, enlargement of palatal tonsils, base of the tongue hypertrophy, visibility of vallecula, pathology of epiglottis), will be performed.

Thereafter, each patient will undergo polysomnography and patients will be divided according to the severity of OSA into three groups (mild OSA - 5 < AHI ≤ 15, moderate OSA 15 < AHI ≤ 25, and severe OSA with AHI > 25 events per hour of sleep).

According to history, otorhinolaryngology examination and polysomnography, presumably site of obstruction will be stated and therapeutic plan will be designated. Patients with severe OSA will be sent for CPAP (continuous positive airway pressure) treatment, whereas surgery will be recommended for patients with mild and moderate OSA.

• Drug-Induced sleep endoscopy

- Indication and contraindication to DISE DISE will be indicated in patients with mild and moderate OSA and in those with severe OSA who will fail or refuse CPAP treatment. All these patients will be potentially planned for surgery and will have to agree with the surgical treatment.

Patients with ASA (American Society of Anesthesiology) score above 4, as well as patients with central apnea and propofol or midazolam allergies, will be excluded from the study.

* Premedication Patients will be pre-medicated with a combination of 5 mg midazolam and 0,5 mg atropine intramuscularly 30 minutes before DISE.
* Procedure Patients will be lying in a supine position on an operation table, the lights will be dimmed and the room quiet to minimize awaking stimuli. Patients will be standardly monitored: ECG (electrocardiogram), blood oxygen saturation, non-invasive blood pressure, and depth of anesthesia will be monitored by bispectral index (BIS). Local anesthesia of nasal cavity will be performed by Lidocaine 10%, 2 sprays into each nostril.

Anaesthesia will be induced by intravenous bolus of propofol 1 mg per kg of ideal body weight, and maintained by repeated boluses of propofol 10-20 mg every 3-5 minutes for the target BIS (Bispectral Index) value of 50-70. Once the patient reaches a satisfactory level of sedation, a flexible fiber optic. Intubation scope 3.7mm x 65cm coated with anti-condense will be introduced into the nasal cavity. The nasal passage, nasopharynx, velum, oropharynx (including tonsils), tongue base, epiglottis, and larynx will be observed. The length of examination will be 15 minutes minimal in order to detect the obstruction. DISE findings will be reported using the VOTE classification system according to Kezirian. Accordingly, localization of upper airways obstructions will be done.

At the end of endoscopy a jaw thrust (or Esmarch maneuver) will be performed. The mandible will be gently advanced up to 5 mm. The manoeuver will be evaluated as successful when the enlargement of upper airway will be observed and disappearance of apnea mimicking the effect of mandibular repositioning appliance (MRA).

After finishing of endoscopy, patients will be awakened to full consciousness in the operating room and then transferred to recovery room for 1-hour observation.

• Evaluation of changes in indication for site of surgery Indication for surgery made according to otorhinolaryngology examination before DISE and after DISE will be compared. Changes will be noted and the number of patients will be calculated using percentage.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years
* obstructive sleep apnoea (mild, moderate Apnea-Hypopnea Index (AHI) <15)
* severe OSA - failed CPAP treatment
* severe OSA - patients whorefused CPAP

Exclusion Criteria:

* ASA 4 (classification of the American Society of Anesthesiologists)
* pregnancy
* propofol or midazolam allergies
* other significant disease with current decompensation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Comparison of indication for surgery based upon ENT examination before and after DISE. | 36 months
  Indication for surgery made according to otorhinolaryngology examination before DISE and after DISE will be compared. There exist a defined number of surgical procedures for which the patient may be indicated, indication for individual surgical procedures will be compared before and after DISE.

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Komínek, prof.MD,PhD,MBA, Study Director — University Hospital Ostrava; Jaroslava Hybášková, MD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aktas O, Erdur O, Cirik AA, Kayhan FT. The role of drug-induced sleep endoscopy in surgical planning for obstructive sleep apnea syndrome. Eur Arch Otorhinolaryngol. 2015 Aug;272(8):2039-43. doi: 10.1007/s00405-014-3162-8. Epub 2014 Jun 28. PMID 24972543
- [Background] Campanini A, Canzi P, De Vito A, Dallan I, Montevecchi F, Vicini C. Awake versus sleep endoscopy: personal experience in 250 OSAHS patients. Acta Otorhinolaryngol Ital. 2010 Apr;30(2):73-7. PMID 20559476
- [Background] Cavaliere M, Russo F, Iemma M. Awake versus drug-induced sleep endoscopy: evaluation of airway obstruction in obstructive sleep apnea/hypopnoea syndrome. Laryngoscope. 2013 Sep;123(9):2315-8. doi: 10.1002/lary.23881. PMID 24167821
- [Background] DE Corso E, Fiorita A, Rizzotto G, Mennuni GF, Meucci D, Giuliani M, Marchese MR, Levantesi L, Della Marca G, Paludetti G, Scarano E. The role of drug-induced sleep endoscopy in the diagnosis and management of obstructive sleep apnoea syndrome: our personal experience. Acta Otorhinolaryngol Ital. 2013 Dec;33(6):405-13. PMID 24376297
- [Background] De Vito A, Carrasco Llatas M, Vanni A, Bosi M, Braghiroli A, Campanini A, de Vries N, Hamans E, Hohenhorst W, Kotecha BT, Maurer J, Montevecchi F, Piccin O, Sorrenti G, Vanderveken OM, Vicini C. European position paper on drug-induced sedation endoscopy (DISE). Sleep Breath. 2014 Sep;18(3):453-65. doi: 10.1007/s11325-014-0989-6. Epub 2014 May 26. PMID 24859484
- [Background] Kezirian EJ, Hohenhorst W, de Vries N. Drug-induced sleep endoscopy: the VOTE classification. Eur Arch Otorhinolaryngol. 2011 Aug;268(8):1233-1236. doi: 10.1007/s00405-011-1633-8. Epub 2011 May 26. PMID 21614467